CLINICAL TRIAL: NCT05289583
Title: Impact of Therapeutic Alliance on Dropout in a Naturalistic Sample of Patients With Borderline Pathology Receiving Residential DBT
Acronym: DBT_dropout2
Status: Completed | Type: Observational
Sponsor: Evangelisches Krankenhaus Bielefeld gGmbH (Other)
Responsible Party: Principal Investigator, Carolin Steuwe, Psych. Psychotherapist, Evangelisches Krankenhaus Bielefeld gGmbH
Other Study IDs: DBT_dropout2
Record Dates: First submitted 2022-03-11; First posted 2022-03-21 (Actual); Last update posted 2022-04-01 (Actual); Status verified 2022-03

CONDITIONS: Borderline Personality Disorder; Psychotherapy; Dropout
MeSH Terms: conditions — Borderline Personality Disorder | interventions — Dialectical Behavior Therapy

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Dialectical Behavior Therapy: The program's purpose is to help patients achieve the following therapeutic goals: (1) reduction of suicidal behaviors, (2) reduction of therapy-interfering behaviors, and (3) other risky or destabilizing behaviors. Standard DBT aims to achieve these goals by (1) conveying behavioral capabilities (skills), (2) motivation for applying these skills, (3) generalization of learned skills to the patient's natural environment, (4) structuring the treatment environment to reinforce functional behavior, and (5) conveying therapeutic resources and motivation to effectively treat patients with BPD.
  Interventions: Behavioral: Dialectical Behavior Therapy

INTERVENTIONS:
Behavioral: Dialectical Behavior Therapy — DBT is a cognitive-behavioral treatment program that was developed to treat suicidal Patients with BPD (Linehan, 1993).

SUMMARY:
Participants with Borderline pathology (≥ 3 DSM-IV-criteria) receiving an inpatient Dialectical Behavior Therapy (DBT) program completed a quality assurance questionnaire set assessing demographic information and pretreatment psychopathology during the days of their inpatient stay. Beyond that, changes of therapists were documented.

ELIGIBILITY:
Inclusion Criteria:

* three or more criteria for BPD as defined by DSM-5 (Borderline Personality characteristics; BPC)

Exclusion Criteria:

* inability to contract and consent,
* other severe mental disorders (bipolar disorder, acute psychosis),
* current alcohol,
* illicit or not prescribed drug use,
* simultaneous participation in other treatment studies,
* pregnancy or breastfeeding,
* an inability to negotiate a non-suicide agreement,
* ongoing traumatic contact with the perpetrator, and
* a Body Mass Index < 16.5.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: For this study, all patients aged from 18 to 65, discharged from our personality disorder inpatient unit between January 2019 and December 2021, and fulfilling three or more criteria for BPD as defined by DSM-IV (Borderline Personality characteristics; BPC) were considered (n = 44).
Sampling Method: Non-Probability Sample
Enrollment: 44 (Actual)
Dates: Start 2019-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-02-28 (Actual)

PRIMARY OUTCOMES:
Rate of Dropout | 8-10 weeks
  premature termination of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Research Department, Bielefeld, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Steuwe C, Berg M, Driessen M, Beblo T. Therapeutic alliance and dropout in patients with borderline pathology receiving residential dialectical behavior therapy. BMC Psychiatry. 2023 Aug 18;23(1):605. doi: 10.1186/s12888-023-05061-8. PMID 37596568